CLINICAL TRIAL: NCT01104350
Title: Phase I Dose-Escalation Study of Image-Guided Radiation Therapy for Bladder-Cancer Patients Undergoing Radiotherapy and Concurrent Gemcitabine Chemotherapy
Brief Title: Image-Guided Radiation Therapy for Bladder-Cancer Patients Undergoing Radiotherapy and Concurrent Gemcitabine Chemotherapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-031
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Bladder Cancer
Keywords: Bladder; Radiotherapy; Gemcitabine; Chemotherapy; 10-031
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine

ARMS (1):
- Radiotherapy and Concurrent Gemcitabine Chemotherapy (Experimental): This is a Phase I dose-escalation study examining the safety and tolerability of intensity modulated external radiation therapy using image-guidance in combination with gemcitabine chemotherapy as an alternative to radical cystectomy.
  Interventions: Other: external radiation therapy with gemcitabine

INTERVENTIONS:
Other: external radiation therapy with gemcitabine — All patients will undergo daily image-guided radiation therapy with concurrent twice weekly gemcitabine chemotherapy. Radiation therapy will begin 2-4 weeks after restaging cystoscopy/fiducial marker placement.
  * Dose level #1: 23.4 Gy/1.8 Gy × 13 fractions (total dose 68.4 Gy)
  * Dose level #2: 27.0 Gy/1.8 Gy × 15 fractions (total dose 72.0 Gy)
  * Dose level #3: 30.6 Gy/1.8 Gy × 17 fractions (total dose 75.6 Gy)

SUMMARY:
The purpose of this study is to test the safety of different amounts (doses) of external radiation therapy (high-energy x-rays that shrink or destroy cancer) combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* MSKCC-reviewed pathologically proven diagnosis of primary bladder urothelial carcinoma without evidence of regional (nodal) or distant spread (cT1-T4a, Nx or N0).
* Karnofsky Performance Scale (KPS) ≥ 70%
* Age ≥18 years old
* Adequately functioning bladder, defined as continent and without the need for an indwelling catheter
* Absolute neutrophil count (ANC) ≥ 1500/mL; platelets ≥ 100,000/mm3 serum bilirubin < 1.5 x the upper limit of normal (ULN); aspartate aminotransferase (AST) and/alanine aminotransferase (ALT) ≤ 1.5 × ULN
* Adequate renal function: calculated creatinine clearance > 30 mL/min/1.73 m2 using the following formula modified Cockcroft and Gault Formula for estimated Creatinine Clearance
* Patients must be considered able to tolerate systemic chemotherapy and pelvic radiation therapy.
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Evidence of distant disease or histologically-proven nodal metastases. Patients with radiologic evidence of lymphadenopathy must have biopsy proof of N0 status.
* Previous pelvic radiation therapy
* Prior systemic chemotherapy non-cisplatin based neoadjuvant for urothelial carcinoma (prior intravesical chemotherapy or immunotherapy is permissible)
* Prior cisplatin based neoadjuvant systemic chemotherapy for more than >4 cycles
* Active inflammatory bowel disease (i.e., Crohn's disease or ulcerative colitis)
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To determine the dose limiting toxicity and establish the maximal tolerated dose | 2 years

SECONDARY OUTCOMES:
To determine the complete response rate of the primary tumor | 4-6 weeks following consolidation therapy
To determine the long term toxicity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Kollmeier, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm